CLINICAL TRIAL: NCT05729165
Title: Local Vibration Therapy and Traditional Speech Therapy for Dysphagia in Patients with Severe Acquired Brain Injury
Brief Title: Local Vibration in Patients with Severe Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, PADUA LUCA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0038189/21
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Acquired Brain Injury; Dysphagia
Keywords: Acquired Brain Injury; Dysphagia; Local vibration; Technological Rehabilitation
MeSH Terms: conditions — Brain Injuries; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Interventional, randomized, parallel assigment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (S-G) (Experimental): 20 minutes of local vibration treatment with the Novafon® Pro medical device followed by 20 minutes of traditional speech therapy, for a total duration of 40 minutes. Therefore, using this instrument, local vibration therapy will be applied at the level of (i) the orbicular muscles of the upper and lower lips, (ii) the masticatory muscles (masseter, temporalis, pterygoid), and (i) local intra-oral and tongue. The Novafon® Pro medical device will be used with the following external and intraoral heads: set senses roller, ball head, disc head, ball head, arrow head, spoon head, and tongue depressor head.
  Traditional speech therapy treatment will be carried out with the same tools and activities already described in the C-G.
  Interventions: Device: Novafon® Pro; Other: Conventional Therapy
- Control group (C-G) (Active Comparator): 40 minutes of conventional speech treatment. Specifically, maneuvers will be performed for (i) extra-oral and intra-oral passive thermal stimulation, (ii) extra-oral and intra-oral passive tactile stimulation, and for (iii) elicitation of active bucco-lingual and laryngeal muscle movements. The following instruments will be used for this purpose: ice cubes, ice tubes, sterile gauze, tongue depressors, swabs, 10 mm laryngeal mirrors.
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Device: Novafon® Pro — Local vibration therapy. The target muscles were: the orbicularis muscles of the upper and lower lips, the masticatory muscles (masseter, temporalis, pterygoidis) and lingual muscles.
  Arms: Experimental group (S-G)
Other: Conventional Therapy — maneuvers were performed for passive extra-oral and intra-oral thermal stimulation, passive extra-oral and intra-oral tactile stimulation, and elicitation of active movements of the bucco-lingual and pharyngo-laryngeal muscles.

SUMMARY:
Severe Acquired Brain Injury (sABI), with a more or less prolonged state of coma, generally causes disruption of the physiological modes of swallowing and feeding and the physiological abilities of communication and phonation.

There is broad agreement in the scientific literature for early intervention by the entire rehabilitation team. In the specific case of swallowing and phonatory function, speech therapist intervention is indicated with the goal of restoring the automatic and voluntary movements of the muscles involved in the performance of the previously mentioned functions.

Speech-language treatment of buccal structures, sensation, motor and praxie is recommended in conjunction with other types of approaches (dietary modifications, compensation techniques, postural modifications).

In the acute and early subacute phase of patients with sABI with a vigilance level of less than 4 according to the Levels of Cognitive Functioning scale, alterations in bucco-linguo-facial structures and swallowing can be observed that prevent the execution of a correct motor pattern of phonation and swallowing. For this reason, passive and/or active stimulation aimed at restoring sensitivity, strength, and movement coordination of the bucco-linguo-facial and laryngeal muscles is necessary to rehabilitate the prerequisites for the initiation of feeding, to restore adequate afferents, and to stimulate communication.

A careful search of the literature shows that over the past decade many studies in the rehabilitation field have sought to understand the effects of local vibration therapy at various levels of the central nervous system and the possible benefits in neurorehabilitation. From a speech therapy perspective, there are only three studies on the area of dysphonia in cases of upper laryngeal nerve palsy, combining traditional treatment with the use of Novafon®, a sound wave medical device used for Local Vibrational Therapy. The results show greater improvements in vocal function and voice quality when classical treatment is combined with Local Vibrational Therapy. These studies conclude by affirming the need for further research with a larger sample size to analyze the potential effectiveness of Novafon® applied to the recovery of vocal cord paralysis.

DETAILED DESCRIPTION:
The purpose of the present study is to observe the effects of integrating traditional speech therapy with the new intervention modality of local vibration therapy with Novafon® in patients with sABI.

Specifically, this study aims to:

(i) Observe and record an increase in trophism of the muscles involved; (ii) improve swallowing and phonatory functions. Twenty-four patients of both sexes with sABI will be recruited, evaluated and treated at the UOC of High Intensity Neurorehabilitation, Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome.

Participants included in the study will be randomized into two groups according to a computer-generated sequence: patients in the experimental group (S-G) will perform traditional speech therapy combined with speech therapy using Novafon®; patients in the conventional group (C-G) will perform only traditional speech therapy.

The experimental rehabilitation treatment will be carried out at the rate of once a day, 5 days a week for a total of 8 weeks. Each speech therapy session will last a total of 40 minutes.

The rehabilitation treatment will be carried out in the room of the patient, who will be placed in a sitting position in a wheelchair or bed, with the backrest inclined at least 45°.

ELIGIBILITY:
Inclusion Criteria:

* Previous coma
* Age between 18 and 90 years
* Level of consciousness greater than or equal to Minimally Conscious State plus
* Feeding through SNG or PEG
* Clinical stability
* Ability of caregiver/legal guardian to understand and sign informed consent

Exclusion Criteria:

- Psychiatric or other conditions that may affect patient compliance with treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Dysphagia Outcome and Severity Scale (DOSS) | Change from baseline DOSS at 4 and 8 weeks
  DOSS is a 7-point functional dysphagia rating scale (from 1 severe dysphagia with the need for artificial feeding, to 7 swallowing in the normal range and exclusive oral feeding), which provides recommendations regarding the type of diet/nutrition to be followed and the level of independence. The progress of this 7-point scale reflects an improvement in the level of dependence in feeding (form 0, "total dependence" to 7, "self-sufficient patient"), level of nutrition (levels 7-3 full oral nutrition and levels 2-1 non-oral nutrition) and type of diet according to different food consistencies (levels 7-6 normal diet consistency, level 5 may need one diet consistency restriction, level 4 one to two diet consistency restrictions, and level 3 two or more diet consistency restrictions). The aspects considered by this scale are bolus management in the oral phase, pharyngeal phase retention and ability to protect the airway.

SECONDARY OUTCOMES:
Bedside Swallow Assessment scale (BSAs) | Change from baseline BSAs at 4 and 8 weeks
  BSAs is a tool with a minimum score of 19 in case of adequate swallowing function and a maximum score of 48 indicating severe discomfort. It is divided into three parts:
  1. level of consciousness, trunk and head control, respiration, structures of the phono-articulatory and swallowing apparatus;
  2. direct evaluation of swallowing by administering 5 ml of water and recording laryngeal movements with attempts to swallow, repetitive movements, the presence or absence of coughing during swallowing and the presence of gurgling voice after swallowing;
  3. administration of 60 ml of water, recording the time required to finish, the number of sips, the presence of coughing, the presence of gurgling voice.
  A scale value < 19 reflects the inability to perform part of the tests, particularly the third part with water administration, due to risk of aspiration, inability or lack of cooperation from the patient.
Fiberoptic Endoscopic Evaluation of Swallowing (FEES) | Change from baseline FEES at 4 and 8 weeks
  FEES is a highly sensitive and useful examination to obtain information on the anatomical rhino-pharyngeal-laryngeal structures, swallowing mechanism, pharyngeal motility, and sensitivity of the pharyngeal-laryngeal tract. FEES does not allow direct verification of whether aspiration is present, but the risk of aspiration can be detected by the presence of post-deglutition stagnation in the laryngeal vestibule.
Phonation | Change from baseline phonation at 4 and 8 weeks
  Phonation will be assessed through the use of a sound level meter, an instrument that can identify the decibels (dB) of phonation.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Padua, MD, phD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No